CLINICAL TRIAL: NCT01080560
Title: A Randomized Single Dose Open Label Bioequivalence Study of Cyclosporine Capsules USP (Modified)100mg in Normal Healthy Male Subjects Under Fasting Condition
Brief Title: Bioequivalence Study of Cyclosporine 100mg Capsule Under Fasting Condition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Panacea Biotec Ltd (Industry)
Responsible Party: Dr. Arani Chatterjee, Panacea Biotec Ltd
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: US/AHD/07/013
Record Dates: First submitted 2010-03-02; First posted 2010-03-04 (Estimated); Last update posted 2010-03-04 (Estimated); Status verified 2010-03

CONDITIONS: Healthy Volunteers
Keywords: Bioequivalence study in healthy volunteers
MeSH Terms: interventions — Cyclosporine; Cyclosporins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- NEORAL® Capsule 100 mg (Active Comparator)
  Interventions: Drug: Cyclosporine Capsules USP (Modified) 100 mg
- Cyclosporine 100 mg Capsule (Experimental)
  Interventions: Drug: Cyclosporine Capsules USP (Modified) 100 mg

INTERVENTIONS:
Drug: Cyclosporine Capsules USP (Modified) 100 mg — Subjects will be administered either Test Product or Reference Product with 240ml of water according to randomization schedule
  Other Names: Cyclosporine Capsule; Gengraf Capsule; Sandimmune Capsule

SUMMARY:
To demonstrate bioequivalence between Test Product (A):Cyclosporine Soft Gelatin Capsules Modified 100 mg manufactured by Panacea Biotec Ltd, India and the corresponding Reference Product (B):Neoral (Cyclosporine capsules,USP)Modified 100mg manufactured by Novartis Pharmaceuticals Corporation, New Jersey, in 36 healthy adult male subjects under fasting condition.

DETAILED DESCRIPTION:
Total 36 normal healthy adult male subjects will be enrolled in the study. Subjects will be administered either the Test or the Reference Product with 240 mL of water in each period as per the randomization schedule. Subjects will fast for at least 10 hours prior to dose administration and for at least 4 hours post dose. Standardized meals will be provided in each study period. Water will not be accessible to the subjects 1 hour Predose and 2 hours Post dose in each period. A total of 24 blood samples will be withdrawn for pharmacokinetic profiling. The whole blood concentrations of Cyclosporine will be measured by a validated LC/MS/MS analytical method. Ratio analysis will be performed for untransformed and log transformed pharmacokinetic parameters Cmax, AUC0-72, AUC0 inf. ANOVA will be performed on log transformed pharmacokinetic parameters Cmax, AUC0-72, AUC0-inf and 90% confidence interval will be constructed for the ratio of geometric least square mean of the Test and Reference products, obtained from the log-transformed data. Bioequivalence will be concluded if the ratio estimate as well as its 90% confidence interval, both falls within the acceptable range of 80.00% to 125.00% for Cmax, AUC0-72 and AUC0-inf.

ELIGIBILITY:
Inclusion Criteria:

1. Male subjects in the range of 18 - 45 years of age.
2. The healthy human subjects, whose body weight within ± 15% of ideal weight as related to height and body frame according to Life Insurance Corporation (LIC) Chart (Appendix A).
3. Subjects with normal findings as determined by baseline history, physical examination and vital signs (blood pressure, pulse rate and body temperature).
4. Subjects with normal findings as determined by hematological tests, Serum Chemistry, serological tests, urine analysis, ECG and X-ray (X-ray if taken).
5. Willingness to follow the protocol requirement as evidenced by written, informed consent.
6. Agreeing to, not using any medication (either prescribed, OTC or alternate medicines), including vitamins and minerals for 14 days prior to study and during the course of the study.
7. No history or presence of significant alcoholism or drug abuse in the past one year.
8. Non-smokers, ex smokers and light smokers will be included. "Light smokers are defined as someone smoking 10 cigarettes or less per day, ex smokers as someone who completely stopped smoking for at least 3 months.

Exclusion Criteria:

1. Requiring medication for any ailment including enzyme-modifying drugs in the previous 28 days, before day one (1).
2. Any medical or surgical conditions, which might significantly interfere with the functioning of gastrointestinal tract, blood-forming organs etc.
3. History of cardiovascular, renal, hepatic, ophthalmic, pulmonary, neurological, metabolic or psychiatric diseases.
4. Subjects with history of recent myocardial infarction, cardiac arrhythmias, cardiac failure and convulsions.
5. Participation in a clinical drug study or bioequivalence study 90 days prior to present study.
6. History of malignancy or other serious diseases.
7. Refusal to abstain from food for at least ten (10.00) hours prior to drug administration and for at least four (04.00) hours post dose.
8. Refusal to abstain from water for at least one (01.00) hour prior to study drug administration on first day of each study period and for at least two (02.00) hours post dose.
9. Any contraindication with blood sampling.
10. Refusal to abstain from smoking or consumption of tobacco products 48.00 hours before dosing until last sample collection of each period.
11. Found positive in Breath alcohol test done at the time of check in for each study period.
12. History of drug abuse in the past one year.
13. Use of xanthine-containing beverages or food, and grape fruit juice for 48.00 hours prior to each drug dose.
14. Blood donation 90 days prior to the commencement of the study.
15. Subjects with positive HBsAg or Hepatitis-C tests or HIV tests or Anti Treponema Palladium/Syphilis test.
16. Known history of hypersensitivity to Cyclosporine or to any component of the formulation.

    -

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2007-08; Primary Completion 2007-09 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
To demonstrate bioequivalence between Test Product,Cyclosporine Soft Gelatin Capsules Modified 100mg of Panacea Biotec and the corresponding Reference Product, Neoral(Cyclosporine Capsule,USP)of Novartis Pharmaceutical Corporation, New Jersey | upto 3 days

SECONDARY OUTCOMES:
To monitor the safety and tolerability in subjects receiving single dose of Cyclosporine Capsule. | upto 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Dr Nirav Gandhi, Principal Investigator — Accutest Research Laboratories (I) Pvt. Ltd.
Locations (1):
- Accutest Research Laboratories (I) Pvt Ltd., Ahmedabad, Gujarat, India